CLINICAL TRIAL: NCT04643418
Title: Phase 1/2a Dose-ranging, Safety, Pharmacokinetics, and Preliminary Efficacy Study of MPB-1734 in Patients With Advanced Solid Tumors in Part 1 and With Selected Solid Tumors in Part 2
Brief Title: Phase 1/2a Study of MPB-1734 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MegaPro Biomedical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DMB-CT-001
Record Dates: First submitted 2020-11-20; First posted 2020-11-25 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Solid Tumor, Unspecified, Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MPB-1734, single arm, dose escalation (Experimental): intravenous, once per 3 weeks, starting at 10 mg/m˄2
  Interventions: Drug: MPB-1734

INTERVENTIONS:
Drug: MPB-1734 — Administered once daily in a 21-day cycle
  Other Names: DMB025

SUMMARY:
This is a first-in-human (FIH), multicenter, open-label, uncontrolled, Phase 1/2a study with dose escalation in patients with advanced solid tumors (Part 1) and cohorts of up to 15 patients per selected indication (Part 2). The solid tumor types in Part 2 will be decided by the sponsor prior to the start of Part 2, but not be solely based on the efficacy results in Part 1.

DETAILED DESCRIPTION:
This study will occur in two parts, Dose-escalation (Part 1) and Cohort-expansion (Part 2). The main purpose of Part 1 is to determine the doses and dosing schedule of MPB-1734 that is safe and tolerable when given in subjects with certain types of advanced cancer. Part 2 of the study will begin when the Sponsor determines the safe and tolerable doses and dosing schedule from Part 1. The main purpose of Part 2 is to continue to assess the safety and tolerability of the MPB-1734 dose and dosing schedule determined by the Sponsor during Part 1. The preliminary efficacy of MPB-1734 will also be assessed in both Part 1 and Part 2.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent in the local language prior to any study-mandated procedure.
2. Male or female patients at least 18 years of age, at the time of informed consent.
3. Male or nonpregnant and nonlactating female patients with pathologically confirmed, measurable solid tumor lesions (Response Evaluation Criteria in Solid Tumors version 1.1 [RECIST 1.1]) that are unresectable, and standard therapy able to provide clinical benefit does not exist or is no longer effective.
4. Eastern Cooperative Oncology Group Performance Status ≤2.
5. Patients have recovered from the acute toxicity of previous therapies (peripheral sensory neuropathy recovered to ≤Grade 2) except alopecia, and:

   * At least 4 weeks have elapsed since completing surgery, endocrine therapy, tyrosine kinase inhibitor therapy, immunotherapy, radiotherapy, chemotherapy, and/or
   * At least 6 weeks have elapsed since completing chemotherapy with nitrosoureas, melphalan, and/or mitomycin C, and/or
   * At least 6 weeks have elapsed since completing cranial radiotherapy.
6. Life expectancy of greater than 12 weeks.
7. Ability to communicate well with the investigator, in the local language, and to understand and comply with the requirements of the study.

Exclusion Criteria:

1. Peripheral sensory neuropathy >Grade 2 (CTCAE version 5.0) at baseline.
2. Patients requiring immediate palliative treatment of any kind including surgery and/or radiotherapy.
3. Serum bilirubin >1.5× ULN.
4. AST and/or ALT >2.5× ULN if no liver involvement, OR AST and/or ALT >5× ULN with liver involvement.
5. Serum creatinine >1.5× ULN, and/or a creatinine clearance of <50 mL/min calculated by Cockcroft Gault.
6. QTc prolongation defined as a QTc with Framingham correction greater than or equal to 470 ms, or significant electrocardiogram (ECG) abnormalities.
7. Known hypersensitivity to taxanes or any excipients of the drug formulation.
8. Female patients who are pregnant, breast-feeding, or planning to become pregnant during the study.
9. Untreated and/or uncontrolled central nervous system metastases.
10. Patients with brain tumors, primary or metastatic.
11. Patients taking concomitant medications anticipated to result in drug-drug interactions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2022-03-08 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation the the maximum tolerated dose(MTD) by safety data | Through the end of the first cycle (Days 1-21).
  Number and incidence of (serious) adverse events (AEs) ([S]AEs), including rate of mild, moderate, and severe hypersensitivity reactions, fluid retention, and sensory neuropathy an adverse event or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first treatment cycle.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergence Adverse Events | Approximately 24 weeks
  Each adverse event will be coded using the Medical Dictionary (version 20.0) system. The severity of the toxicities will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (version 4.0).
Maximum observed plasma concentration (Cmax) | Day 1-Day 2
  Evaluation the change of Cmax
Area under the plasma concentration-time curve (AUC) | Day 1-Day 2
  Evaluation the change of AUC
Half-life (T1/2) | Day 1-Day 2
  Evaluation of T1/2

CONTACTS AND LOCATIONS:
Overall Officials: Muh-Hwa Yang, MD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No